CLINICAL TRIAL: NCT06673875
Title: Assessment of Pelvic Floor Muscle Training Using Modern Conservative Methods in the Therapy of Stress Urinary Incontinence
Acronym: Aniball-inco
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Martina Szypulova, Doctor of Medicine, gynecologist, urogynecologist, principal investigator, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aniball inco
Record Dates: First submitted 2024-09-14; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; physiotherapy of pelvic floor; conservative treatment
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aniball-inco (Experimental): training muscles with vaginal device to excercise of pelvic floor muscle.
  Interventions: Device: vaginal device Aniball INCO
- RHB (Active Comparator): training muscles without device to excercise of pelvic floor muscle.
  Interventions: Procedure: conservative treatment of stress urinary incontinence - pelvic floor muscle training

INTERVENTIONS:
Procedure: conservative treatment of stress urinary incontinence - pelvic floor muscle training — evaluation of pelvic floor muscle rehabilitation to change the clinical severity of urinary incontinence
  Arms: RHB
Device: vaginal device Aniball INCO — the firt group - the pelvic floor muscle training with vaginal device Aniball INCO according manual after education by the urogynecologist, who is educated in pelvic floor dysfunction.
  the second group - the pelvic floor muscle training without vaginal device, the education was performed by certified physiotherapist trained in pelvic floor disorder.
  Arms: Aniball-inco

SUMMARY:
The eim is to evaluate the clinical effectiveness of pelvic floor muscle training (PFMT) in conservative therapy in women with objective, urodynamic stress urinary incontinence using home exercise training with the medical vaginal device versus standard pelvic floor muscle training-exercises

DETAILED DESCRIPTION:
The first group were using vaginal device - commercial name Aniball INCO®, which is controlled by the Czech State Institute of Drug Control which is registered by the European Medical Device Nomenclature (EMDN) with Unique Device Identifier - Device Identifier (UDI-DI) - 859418371002LA

The second group - the education was provided by certified physiotherapist trained in pelvic floor disroder

ELIGIBILITY:
Inclusion Criteria: stress urinary incontinence

Exclusion Criteria: age under 18, age over 80, ISD (Intrinsic Sphincter Deficiency), descent of the pelvic organs according to POP-Q ≥ 2 (stage), urgent incontinence ruled out using a questionnaire (OAB V8 - overactive bladder < 7a PPIUS - patient perception of intensity and urgency scale ≤ 1), overactive bladder (OAB) with the use of anticholinergics, pregnant women and women up to 6 months after childbirth, active pelvic cancer, degenerative neurological or myofascial disease, reduced cognitive function that does not allow understanding the principles of the study, impossibility of contraction mm.levatores ani., recurrent vaginal inflammation, atrophic vulvovaginitis, irregular bleeding, contraindications listed by the manufacturer of the medical device Aniball inco.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire - urinary incontinence short form (ICIQ-SF) questionnaire | baseline at time of initial urogynecology examination/ after 8 weeks/ and after 4 months at output urogynecology examination
  Assessment of pelvic floor muscle rehabilitation training to change the clinical severity of urinary incontinence using the questionnaire - International Consultation on Incontinence Questionnaire - urinary incontinence short form (ICIQ-UI SF - range 0 to 21) at at time of initial urogynecology examination / after 8 weaks of training / and after 4 months of training/ at the time of output urogynecology examination - in the group with home exercises using the medical device Aniball-inco ( 1st group) vs. exercise of the pelvic floor muscles after education by a physiotherapist (2nd group).

SECONDARY OUTCOMES:
objective urodynamics parameters | baseline at time of initial urogynecologic check visit/ after 4 months at time of output urogynecology examination
  evaluation of changes in urodynamic parameters before pelvic floor muscle training at at time of initial urogynecology examination and after 4 months of training at the time of output urogynecology examination. We will assess the rate of maximum urethral closure pressure (MUCP cmH2O) in two monitored groups.
objective measured parameters of urine leakage. | baseline at time of initial urogynecologic check visit/ after 4 months at time of output urogynecology examination
  Evaluation of the rate of urine leakage using a one-hour pad-weight test (grams). The test is standardised by ICS (International Continence Society).
  The total amount of urine leaked is determined by weighing the pad. The test is performed before training before pelvic floor muscle training at time of initial urogynecology examination and after 4 months of training at the time of output urogynecology examination.

OTHER OUTCOMES:
Ultrasound parameters | baseline at time of urogynecologic check visit/ after 4 months at time of output urogynecology examination
  Ultrasound parameters are evaluated at the time of input urogynecology examination before training and after finishing the study. Parameters are: The mobility of the ureterovesical junction - lines h (millimetr). Gamma angle rotation (°) of urethra. Line p (mm) - diameter of line urethrovesical junction and caudal point of symphysis pubis. Changes in the area of the genital hiatus (Genital hiatus/Genital hiatus volume) - values in square centimetr. Every parameter was measered at rest and at maximum Valsalva manevr. It will be measered before training at time of initial urogynecology examination and after finishing training at time of output urogynecology examination. These will be evaluated as optional tertiary parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Szypulova, Principal Investigator — Investigator
Locations (1):
- University Hospital Brno, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
after enrollment and finishing the study, we will share the data of our research analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2025